CLINICAL TRIAL: NCT00217607
Title: Multicentric Phase II Study Evaluating the Efficacy and Toxicity of Weekly Paclitaxel in Locally Advanced or Metastatic Soft Tissue Angiosarcomas That Cannot be Treated by Surgery
Brief Title: Paclitaxel in Treating Patients With Locally Advanced or Metastatic Soft Tissue Angiosarcoma or Lymphangiosarcoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441642; FRE-FNCLCC-SARCOME-06/0409; EU-20517
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Sarcoma
Keywords: adult angiosarcoma; recurrent adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel (Experimental): Paclitaxel 80 mg/m² Day 1, Day 8 and Day 15. No treatment on Day 22.
  1 cycle = 28 days.
  Treatment duration: 6 cycles (=6 months)
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well paclitaxel works in treating patients with locally advanced or metastatic soft tissue angiosarcoma or lymphangiosarcoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 2-month objective response rate in patients with locally advanced or metastatic, unresectable soft tissue angiosarcoma or lymphangiosarcoma treated with paclitaxel.

Secondary

* Determine the 4- and 6-month response rate in patients treated with this drug.
* Determine tolerability of this drug in these patients.
* Determine the time to disease progression and overall survival of patients treated with this drug.
* Determine the clinical criteria predicting response in patients treated with this drug.
* Correlate the efficacy of this drug with the expression of genes involved in angiogenesis regulation in these patients.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue angiosarcoma or lymphangiosarcoma

  * Locally advanced or metastatic disease
  * Unresectable disease
* Angiosarcomas in previously irradiated areas allowed provided disease is clearly progressive
* Measurable disease
* No Kaposi's sarcoma

PATIENT CHARACTERISTICS:

Age

* 18 to 70

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin < 3 times upper limit of normal (ULN)
* SGOT and SGPT < 2.5 times ULN
* No severe liver failure

Renal

* Creatinine clearance > 60 mL/min
* No severe kidney failure

Cardiovascular

* LVEF ≥ 50%

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No weight loss ≥ 20% of body weight prior to illness
* Patient must be amenable to receiving care during the day
* No HIV positivity
* No clinical neuropathy
* No known allergy to study drug or to any of its components (e.g., Cremophor EL)
* No other progressive malignant tumor
* No chronic illness (somatic or psychiatric) that would preclude study compliance and follow-up
* No psychological, geographical, or social reason that would preclude study follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 2 prior courses of chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Other

* No other concurrent anticancer therapy
* No concurrent participation in another therapeutic investigational study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2008-04 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 2 months

SECONDARY OUTCOMES:
Response rate | 4 months
Response rate | 6 months
Tolerability | 6 months
Time to progression | 5 years
Overall survival | 5 years
Clinical criteria predicting response | 2 months
Correlation of efficacy with the expression of genes involved in the angiogenesis regulation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Penel, MD, Study Chair — Centre Oscar Lambret
Locations (23):
- France (23):
  - Centre Paul Papin, Angers
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot - Lyon, Lyon
  - CHU de la Timone, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - Institut Curie Hopital, Paris
  - Hopital Cochin, Paris
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared at an individual level.

REFERENCES:
- [Result] Penel N, Bui BN, Bay JO, Cupissol D, Ray-Coquard I, Piperno-Neumann S, Kerbrat P, Fournier C, Taieb S, Jimenez M, Isambert N, Peyrade F, Chevreau C, Bompas E, Brain EG, Blay JY. Phase II trial of weekly paclitaxel for unresectable angiosarcoma: the ANGIOTAX Study. J Clin Oncol. 2008 Nov 10;26(32):5269-74. doi: 10.1200/JCO.2008.17.3146. Epub 2008 Sep 22. PMID 18809609